CLINICAL TRIAL: NCT01843439
Title: Effects of Multidisciplinary Interventions in Elderly Asthma Patients With Risk of Acute Exacerbation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sang-Heon Cho (Other)
Collaborators: Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor-Investigator, Sang-Heon Cho, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-1205-083-410
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Asthma; Aged
Keywords: Acute exacerbation; Quality of life; Magnesium deficiency; Multidisciplinary intervention
MeSH Terms: conditions — Asthma; Magnesium Deficiency | interventions — Magnesium; Vitamin B 6; Educational Status; Hotlines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): We designed a intervention study to correct additional risk factors in elderly asthma patients.
  We offer following specific interventions simultaneously to intervention arm and will measure the effects of interventions after 1 years.
  1. popularize and educate the asthma action plan
  2. run a emergency call system for acute exacerbation
  3. educate the proper techniques using inhalers
  4. correct the deficiency of magnesium (magnesium 500mg per day)
  Interventions: Dietary Supplement: Magnesium; Behavioral: Education for asthma action plan; Behavioral: hot-lines for acute exacerbation of asthma; Behavioral: Inhaler technique training

INTERVENTIONS:
Dietary Supplement: Magnesium
  Other Names: Product name - Magnes; Composition - Magnesium Lactate 470mg, Pyridoxine HCl 5mg; Company - Daewha pharmaceutical
Behavioral: Education for asthma action plan
Behavioral: hot-lines for acute exacerbation of asthma
Behavioral: Inhaler technique training

SUMMARY:
We want to examine the effect of multidisciplinary interventions in asthma patients who had experienced acute exacerbation of asthma.

In our previous observational studies, elderly asthma patients had a some distinct features such as impairment of cognitive function, deficiency of micronutrient and absence of caregiver compared with young adult asthmatics.

We wanted to evaluate whether the long-term course of asthma could be modified by intervening deficienies which were found in elderly patiensts.

So, we designed a interventional study to correct above risk factors in elderly asthma patients, which could be aggravating their asthma. Followings are our specific multidiciplinary items that we want to correct.

1. popularize and educate the asthma action plan
2. run a emergency call system for acute exacerbation
3. educate the proper techniques using inhalers
4. correct the deficiency of magnesium (magnesium 500 mg per day)

After 1 years, we will measure the numbers of acute exacerbations, lung function including FEV1 and FEV1/FVC, health-related quality of life and level of serum magnesium in study patients.

ELIGIBILITY:
Inclusion Criteria:

* elderly asthma patients who had experienced acute exacerbation of asthma

  1)aggravations of any of major criteria
* dyspnea
* cough
* wheezing
* increase or purulent changes of sputum
* nocturnal symptoms

  2)aggravation of more than one of following criteria
* a reduction of forced expiratory volume at one second or peak expiratory flow rate more than 20% compared than one's best score
* unscheduled clinic or emergency department visit or admission
* step-up of dose of asthma medications or any intake of systemic steroids

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 360 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Number of acute exacerbation of asthma | 1 year from enrollment
  measure the existence of acute exacerbation when they visit the clinic at 3, 6, 12 month after enrollment

SECONDARY OUTCOMES:
Pulmonary function test | 1 year after enrollment
  measure when subjects visits the clinic at 3, 6, 12 month after enrollment
Asthma control status | one year from enrollment
  measure when subjects visit the clinic at 3, 6, 12 month after enrollment
asthma quality of life questionnaire | one year from enrollment
  measure when subjects visit the clinic at 3, 6, 12 month after enrollment
serum magnesium level | one year from enrollment
  measure when subjects visit the clinic at 3, 6, 12 month after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Heon Cho, MD./PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea